CLINICAL TRIAL: NCT01414088
Title: The Effects of Isotonic and Hypertonic Saline Infusion on Renal Biomarkers for the Measurement of Sodium and Water Channel Activity in the Nephron in Healthy Young Subjects
Brief Title: The Effects of Isotonic and Hypertonic Saline Infusion on Renal Biomarkers in Healthy Young Subjects
Acronym: NARA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: Principal Investigator, Erling Bjerregaard Pedersen, DMSc, Regional Hospital Holstebro
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: EBP-JMJ-2011-1
Record Dates: First submitted 2011-08-09; First posted 2011-08-11 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Nephropathy
Keywords: Nephrology; ENaC; NCC; NKCC; Sodium channels; renal biomarkers
MeSH Terms: conditions — Kidney Diseases | interventions — Sodium Chloride; Saline Solution, Hypertonic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- glucose (Placebo Comparator): glucose 5 %
  Interventions: Other: glucose 5%
- isotonic saline (Active Comparator): isotonic saline 0.9 mg/ml
  Interventions: Other: isotonic saline 0,9 mg/ml
- hypertonic saline (Active Comparator): hypertonic saline 2.9 mg/ml
  Interventions: Other: hypertonic saline 2,9 mg/ml

INTERVENTIONS:
Other: isotonic saline 0,9 mg/ml — infusion, 23 ml/kg, during 50 minutes
  Other Names: isotonic saline
  Arms: isotonic saline
Other: hypertonic saline 2,9 mg/ml — infusion, 7 ml/kg, during 50 minutes
  Other Names: hypertonic saline
  Arms: hypertonic saline
Other: glucose 5% — infusion, 23 ml/kg, during 50 minutes
  Other Names: glucose 5 %
  Arms: glucose

SUMMARY:
The kidneys have numerous salt and water channels and play a major role in the regulation of sodium and water. We do not know how these channels work in certain water and sodium accumulating medical conditions.

The purpose of this study is to identify and measure the activity in the water and sodium channels by measuring urine biomarkers/proteins in young healthy subjects.

DETAILED DESCRIPTION:
25 healthy subjects from age 18-45 are recruited.

Subjects will be examined on three examination days. Four days prior to the examination days the subjects will consume a standard diet based on the amount of sodium and calories.

On the examination day subjects are randomised to an infusion with either isotonic saline 23 ml/kg, hypertonic saline 7 ml/kg or glucose 23 ml/kg for a period of 50 minutes.

Renal function is measured by renal clearance of 51Cr-EDTA, urinary sodium, potassium and creatinine.

Urinary NCC, NKCC and ENAC will be measured to evaluate the activity of sodium channels in the nephron.

ELIGIBILITY:
Inclusion Criteria:

* healthy males and females
* age 18-45
* BMI range 18,5-30,0 kg/m2

Exclusion Criteria:

* hypertension (ie ambulatory BP >130 mmHg systolic or/and >80 mmHg diastolic)
* history or clinical significant signs of heart, lung, liver, kidney, endocrine, brain or neoplastic disease.
* alcohol abuse
* drug abuse
* smoking
* pregnancy or nursing
* blood donation within a month prior to examination
* Medical treatment apart from oral contraception

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2011-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Renal biomarkers | day one
  Urinary epithelial sodium channels (ENaC), Sodium-Chloride transporters (NCC), Sodium-potassium-2chloride transporters (NKCC) and aquaporin2 channels (AQP2) before, during and after fluid infusion

SECONDARY OUTCOMES:
blood hormones regulating salt, water and blood pressure | day one
  plasma concentrations of: renin, Angiotensin II, Vasopressin, atrial natriuretic peptide (ANP) and brain natriuretic peptide (BNP)

CONTACTS AND LOCATIONS:
Overall Officials: Erling B Pedersen, Professor, Study Director — Medicinsk Forskning, Regionshospitalet i Holstebro
Locations (1):
- Medicinsk Forskning, Regionshospitalet i Holstebro, Holstebro, Denmark

REFERENCES:
- [Derived] Jensen JM, Mose FH, Bech JN, Nielsen S, Pedersen EB. Effect of volume expansion with hypertonic- and isotonic saline and isotonic glucose on sodium and water transport in the principal cells in the kidney. BMC Nephrol. 2013 Sep 26;14:202. doi: 10.1186/1471-2369-14-202. PMID 24067081